CLINICAL TRIAL: NCT00315835
Title: A Single Dose, Randomized, Double-Blind, Parallel Group Study of the Safety and Pharmacokinetics of Buprenorphine TDS (12.5, 25, 50 Mcg/Hour) Vs. Placebo in Patients With Moderate to Severe Pain Following Orthopedic Surgery
Brief Title: Safety of the Buprenorphine Transdermal Delivery System in Subjects With Mod-to-Sev Pain Following Orthopedic Surgery.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP96-0104
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2006-04-19 (Estimated); Status verified 2006-04

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; opioid; transdermal
MeSH Terms: conditions — Pain, Postoperative

INTERVENTIONS:
Drug: Buprenorphine transdermal delivery system

SUMMARY:
The objective of this study is to assess the safety of the buprenorphine transdermal system (5, 10, and 20 mg) in comparison to placebo transdermal system in subjects with moderate to severe pain after orthopedic surgery. The double-blind treatment intervention duration is 72 hours during which time supplemental analgesic medication (intravenous morphine PCA) will be provided to all subjects in addition to study drug.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over twenty-five years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain. Transdermal systems may offer advantages over currently indicated oral products including ease and convenience of use, improved compliance, possible reduction in patient care, and prolonged and consistent delivery of drug.

ELIGIBILITY:
Inclusion Criteria:

* underwent any major orthopedic surgical procedure requiring general anesthesia, and were expected to be hospitalized >/=4 days postoperatively.
* in moderate or greater pain post-recovery from anesthesia and were expected to be in, or greater than, moderate pain, without analgesics, for >/=4 days post-surgery.

Exclusion Criteria:

* receiving chronic opioid therapy preoperatively for >1 month that was at a total daily dose of >/= 60 mg of oral morphine equivalents.
* have significant concurrent pulmonary conditions.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1996-10; Study Completion 1997-11

PRIMARY OUTCOMES:
clinical laboratory tests
vital signs
physical examinations
electrocardiograms
elicited opioid side effects
pulmonary function tests (O2 saturation, peak flow, forced expiratory volume, forced vital capacity, respiratory rate, and respiratory depression/hypoxia)
adverse events
application site skin observations
plasma concentrations of buprenorphine at hours 0, 2, 4, 6, 12, 24, 30, 36, 48, 54, 60, 72, 78, or at early termination

SECONDARY OUTCOMES:
pain intensity
acceptability of therapy
quality of sleep
rescue dose usage

CONTACTS AND LOCATIONS:
Locations (1):
- Park Place Therapeutic Center, Plantation, Florida, United States